CLINICAL TRIAL: NCT04385264
Title: #StayHome: Efficacy of Early Hydroxychloroquine in Outpatients to Reduce Secondary Hospitalisation and Household Transmission of COVID-19 in Switzerland: A Double-blind, Randomised, Placebo-controlled Trial
Brief Title: #StayHome: Early Hydroxychloroquine to Reduce Secondary Hospitalisation and Household Transmission in COVID-19
Acronym: #StayHome
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sufficient number of subjects would probably not reach
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Unisante
Record Dates: First submitted 2020-04-21; First posted 2020-05-12 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (Mannitol), oral capsules Day 0: 4 capsules PO OD Days 1-5: 2 capsules PO OD
  Interventions: Drug: Mannitol
- Hydroxychloroquine (Experimental): Hydroxychloroquine 200mg (HCQ, Plaquenil), oral capsules Day 0: 800mg PO OD (4 capsules) Days 1-5: 400mg PO OD (2 capsules daily)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Day 0: 800mg PO OD (4 capsules) Days 1-5: 400mg PO OD (2 capsules daily)
  Other Names: Plaquenil; HCQ
  Arms: Hydroxychloroquine
Drug: Mannitol — Day 0: 4 capsules PO OD Days 1-5: 2 capsules daily PO OD
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
BACKGROUND Despite drastic quarantine measures, COVID-19 continues to propagate and threatens global healthcare systems by saturating their capacity with high transmissibility and the particularly protracted length of stay needed by those requiring intensive care. Indeed, once patients advance to the ICU, prognosis is poor and it is thus critical to test medications that may prevent complications and reduce viral shedding. i.e. to protect ambulatory patients and their families from complications and transmission and allow them to #StayHome.

To date, no treatment has been reliably demonstrated as effective in COVID-19 patients.

Hydroxychloroquine (HCQ), a common and well tolerated medication, has shown promise in vitro for reducing viral replication (for SARS-CoV-2 as well as other coronaviruses with pandemic potential such as SARS-CoV-1 and MERS). Since then, several small-scale hospital-based clinical studies have indicated the potential for reduced viral shedding and hospitalisation as well as favourable evolution of lung pathology. If started earlier, this treatment could prevent complications requiring hospitalisation and intensive care, which may not be available in low-income countries.

Robust clinical trials are required to assess the potential of HCQ in COVID-19.

OBJECTIVES This trial assesses the efficacy of early treatment with HCQ in COVID-19 outpatients to reduce the incidence and severity of complications including secondary hospitalisation, ICU admissions, lung pathology and death. Secondarily, this trial will also assess its efficacy to reduce viral transmission among household contacts during self-quarantine. The clinical data collected in this trial will also be critical in creating early prognostication models to better predict healthcare needs and have evidence-based prioritization of resource allocation, which is especially critical in low-resource settings.

METHODS The trial will recruit 800 SARS-CoV-2+ patients and their household contacts at triage sites across Switzerland. Patients included are 1) at risk of poor outcome (comorbidities or >65y) and 2) well enough to self-isolate at home. These patients will be randomised 1:1 in HCQ:Placebo and given 6 days of early treatment (within 24 hours of the SARS-CoV-2 test). Intensive pragmatic multiparameter at-home follow-up (including point-of-care lung ultrasound in some sites) will continue until their outcome (resolution, or complications, such as hospitalisation, ICU admission, death). Household contacts will have before and after serological testing and social distancing knowledge and practices questionnaires to assess risk factors for infections. The household attack rate of new-onset infections can then assess the efficacy of HCQ to prevent transmission.

ELIGIBILITY:
INCLUSION CRITERIA (index cases):

* Age >=18 years old AND
* SARS-CoV-2 positive AND
* Well enough to self-isolate at home (at an address in Switzerland) AND
* At risk of complications from COVID-19 i.e. one or more of the following

  * Age >=65 years
  * Hypertension
  * Diabetes
  * Cardiovascular disease (History of infarction OR peripheral arteriopathy OR cerebrovascular accident OR cardiac insufficiency)
  * Chronic respiratory disease
  * Immunosuppression
  * Cancer
  * Obesity (BMI>40)

EXCLUSION CRITERIA (index cases):

* Allergy to hydroxychloroquine/4-aminoquinilones
* Retinal eye disease
* Known chronic kidney disease, stage 4 or 5 or receiving dialysis
* Weight < 40 kg
* Known porphyria
* Known psoriasis
* Known myasthenia gravis
* Taking drugs with moderate-severe interactions with HCQ
* Taking ≥ 2 QT prolonging drugs
* Taking 1 QT prolonging drug AND a loop diuretic
* Moderate or severe heart failure
* Severe or uncontrolled arrhythmia
* Recent myocardial infarction or stroke (past 6 months)
* Current pregnancy
* Current hospitalisation
* Known hemolytic anaemia

INCLUSION CRITERIA (household contacts):

* Age >1 year old AND
* Living in same household as index case during self-isolation

EXCLUSION CRITERIA (household contacts):

* History of laboratory-confirmed SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of poor outcomes (in index cases) | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  Proportion of secondary hospitalisations (and their length), ICU admissions (and their length) and deaths.

SECONDARY OUTCOMES:
Secondary household attack rate (in household contacts) | From day 0 (diagnosis and enrolment of index case) to 14 days after the outcome of the index case is recorded (recovery, hospitalisation or death): Average of 25 days
  Proportion of a household with new seropositivity for SARS-CoV-2
Subjective disease severity (in index cases) | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  An ordinal scale of disease severity using a visual analogue scale (0-10 where 0 is asymptomatic)
Rate of acute respiratory distress syndrome (in index cases) | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  As recorded during hospitalisation
Severity of radiological lung pathology (in index cases) | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  Measured with lung ultrasound, CT or x-ray
Objective disease severity (in index cases) | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  An ordinal scale of disease severity using the evolution of clinical biomarkers such as oxygen saturation, respiration rate etc.
Safety: Unintended toxic HCQ accumulation (in index cases) | During the period that the subject is considered as COVID-19-positive : Average of 11 days
  Plasma concentrations of HCQ measured by liquid chromatography-tandem mass spectrometry
Safety: Adverse events (in index cases) | During the period that the subject is considered as COVID-19-positive : Average of 11 days
  Ambulatory ECG and intensive monitoring for adverse events
Social distancing knowledge, attitudes and practices amongst index cases and household contacts | During the period that the subject is considered as COVID-19-positive: Average of 11 days
  Visual analogue scores for social distancing practices (0-5, where 0 is no social distancing at all)

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD-PhD, Principal Investigator — Unisanté; Mary-Anne Hartley, MD, PhD MPH, Principal Investigator — Unisanté
Locations (1):
- Unisanté, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The aim is to share data, protocols, information sheets, CRFs and analytical code as soon as possible. Data will first be cleaned and anonymised and then subjected to rigorous assessments to secure patient privacy and analytical robustness according to the FAIR principles.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Unknown (determined by the evolution of the epidemic)
Access Criteria: On request by researchers agreeing to use the data for it intended purpose: i.e. to further knowledge of the efficacy and safety of HCQ in COVID-19 and to better understand the disease.